CLINICAL TRIAL: NCT01284036
Title: Ascending Single Dose Study Of The Safety, Tolerability, And Pharmacokinetics Of PF-05230905 Administered Subcutaneously Or Intravenously To Healthy Subjects
Brief Title: A Single Dose Study Of The Safety And Investigational Product Level Measurement In Healthy Subjects
Acronym: FIH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple
Other Study IDs: B2331001; 3294K1-1000
Record Dates: First submitted 2010-09-29; First posted 2011-01-26 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: Healthy subject; safety; PK study; healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-05230905 (Other): 9 subjects will participate in each dose cohort. 6 subjects will receive investigational product (PF-05230905) and 3 subjects will receive placebo
  Interventions: Drug: PF-05230905

INTERVENTIONS:
Drug: PF-05230905 — Single dose subcutaneous or intravenous (IV) administration of PF-05230905 or placebo

SUMMARY:
The purpose of this study is to find the safety and side effects of investigational drug in healthy volunteers. See how quickly investigational drug enters the bloodstream, is distributed in the body, broken down and removed in healthy male and female volunteers. See if your body makes antibodies to this investigational drug (how your immune system responds).

DETAILED DESCRIPTION:
First in human study to collect safety and pharmacokinetics (PK) of single ascending dose in Healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication.
* Receipt or treatment with an investigational or marketed biologic drug.
* blood donation of approximately 1 pint (500 mL) within 56 days prior to dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2010-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Safety endpoints will be evaluated by comparing reported adverse events in subjects receiving PF-05230905 versus subjects receiving placebo. | day 168
Incidence and severity of clinical laboratories including absolute hepatic transaminases and bilirubin levels will be evaluated. | day 168
Mean change from baseline in vital signs measurements. Mean change from baseline in 12 lead echocardiogram (ECG) will be compared to ensure safety of the subjects. | day 168

SECONDARY OUTCOMES:
Incidence of development of Anti Drug Antibody. | day 168
Serum PF-05230905 concentrations will be determined by a validated assay, and noncompartmental pharmacokinetics (PK) parameters. | day 168
Urine pharmacokinetics (PK) parameters amount excreted in urine (Ae) and renal clearance will be determined. | day 168

CONTACTS AND LOCATIONS:
Overall Officials: Josefin-Beate Holz, MD, Study Director — Ablynx, a Sanofi company
Locations (1):
- Investigational Site, Tacoma, Washington, United States